CLINICAL TRIAL: NCT04361214
Title: Leflunomide for the Treatment of Ambulatory Patients With Mild COVID-19
Brief Title: Leflunomide in Mild COVID-19 Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by PI
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0622
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: leflunomide
MeSH Terms: conditions — COVID-19 | interventions — Leflunomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Leflunomide (Experimental): Leflunomide 300 mg once daily administered for three days followed by 30 mg once daily administered for two days or until fevers abate (maximum ten days of treatment allowed).
  If patients report symptoms attributed to the medication, the dose will be administered at 50 mg once daily for the loading dose followed by 20 mg once daily.
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — Tolerability study of leflunomide 100 mg administered once daily for 3 days followed by 30 mg administered once daily for the duration of 2 - 7 days.

SUMMARY:
This study aims to examine the tolerability of high dose of leflunomide in patients with COVID-19 who are being managed in the outpatient setting.

DETAILED DESCRIPTION:
This is a single are and single-center tolerability study of high dose leflunomide therapy in outpatient adult participants with mild COVID-19. In vitro studies have shown antiviral effects of leflunomide against SARS CoV-2, but the clinical outcomes in the disease have been variable. Our hypothesis is that targeting high risk patients earlier in the disease course and with a higher dose regimen are both required to see improvement in disease outcome measures in COVID-19. This study aims to prove the tolerability of high dose leflunomide in this setting.

Patients are selected based on identification of mild COVID-19 symptoms. Investigators will enroll twenty patients and perform a detailed Tele-helath interview to ensure they meet eligibility criteria and provide informed consent. 100 mg leflunomide daily for three days followed by 30 mg day will be prescribed. The subjects will be required to monitor their temperatures twice daily and a daily telephone call with an investigatory will review symptoms of disease and potential side effects of the drug. Subjects can discontinue the drug after five days if they no longer have fever, or take the drug for up to ten days if required for fever resolution.

ELIGIBILITY:
Inclusion Criteria:

* Being tested positive for SARS-Cov-2 in outpatient setting in drive-thru, ED, or ambulatory clinics at the University of Chicago within 72 hours of enrollment.
* Age >18
* Mild COVID-19, defined as the presence of any symptom consistent with an upper respiratory tract infection, including dry cough, sore throat, nasal congestion, fatigue, myalgia, headaches

Exclusion Criteria:

* Participation in any other clinical trial of an experimental agent treatment for COVID-19
* Current hospitalization
* Known hypersensitivity to leflunomide
* Currently taking methotrexate
* Currently taking terliflunomide
* Known chronic kidney disease, stage 4-5, or receiving dialysis
* History of liver disease
* History of interstitial lung disease
* Pregnancy and lactation - pregnancy test required for females
* Inability to monitor body temperature (oral, axillary, tympanic or frontal) at least twice a day from study enrollment day (Day 1) to the end of the study (Day 14).
* Inability to provide informed consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Tolerability of high dose leflunomide as measured by leflunomide dose modifications | 14 days
  Number of subjects requiring leflunomide dose modifications
Tolerability of high dose leflunomide as measured by discontinuation of leflunomide | 14 days
  Number of subjects that discontinue leflunomide
Tolerability of high dose leflunomide as measured by Adverse Events | 14 days
  Number of Adverse Events observed in all subjects for the duration of the study

SECONDARY OUTCOMES:
Time to defervescence as measured in days while on treatment protocol | 14 days
  The number of days to reach first fever normalization (criteria for normalization: temperature < 100.4 F)
Resolution of other COVID-19 symptoms measured in days while on treatment protocol | 14 days
  Number of days to resolve other symptoms, as assessed by a standardized questionnaire for symptom assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millis, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No